CLINICAL TRIAL: NCT05467761
Title: A Phase 1 Study Comparing the Pharmacokinetics and Safety of Intravenous and Oral Psilocybin
Brief Title: Bioavailability Study of Psilocybin in Normal Adults
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor was not financially able or willing to continue to support the study
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: TRYP Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2022-0612; A561000 (Other: UW Madison); PHARM/PHARMACY (Other: UW Madison); 04/21/2022 (Other: UW Madison); 2022-0612 (Other: UW Madison)
Record Dates: First submitted 2022-07-18; First posted 2022-07-20 (Actual); Last update posted 2023-05-15 (Actual); Status verified 2023-05

CONDITIONS: Healthy
Keywords: psilocybin; psychedelics
MeSH Terms: interventions — Psilocybin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Oral and IV psilocybin (Experimental): Psilocybin with psychological support: Psilocybin will be administered in the form of capsules, taken orally with water, at one visit. Psilocybin will be administered through IV at the other visit.
  Interventions: Drug: Oral Psilocybin; Drug: IV Psilocybin

INTERVENTIONS:
Drug: Oral Psilocybin — 25mg orally
Drug: IV Psilocybin — 5mg intravenously

SUMMARY:
The purpose of this research study is to compare an oral dose of psilocybin and an intravenous (IV) infusion of psilocybin to assess differences in how the drug is absorbed by the body, the psychedelic experience, and any side effects when taken by healthy adult participants. Participants can expect to be in the study for approximately 12 weeks.

DETAILED DESCRIPTION:
Psilocybin, when delivered to screened and prepared participants in a controlled environment, has shown strong evidence of positive effects in treating cancer-related psychiatric distress, depression and anxiety, treatment-resistant depression, and nicotine or alcohol addiction. Psilocybin therapy is generally safe and well-tolerated when conducted under controlled conditions. Psilocybin is very rapidly transformed to the active metabolite psilocin, which is considered the active agent from psilocybin administration. Oral and IV psilocybin are expected to have similar pharmacokinetic and psychedelic effects, as well as safety profiles, while IV psilocybin will achieve more consistent blood levels than are possible with oral psilocybin.

ELIGIBILITY:
Inclusion Criteria:

* Overall healthy and medically stable, as determined by screening
* Capable of giving signed informed consent
* Negative urine pregnancy test in persons of childbearing potential

Exclusion Criteria:

* Have any of the following cardiovascular conditions: uncontrolled hypertension, coronary artery disease, congenital long QT syndrome, cardiac hypertrophy, cardiac ischemia, congestive heart failure, prior myocardial infarction, tachycardia, artificial heart valve, corrected QT interval (QTc) >450 msec at screening, any other clinically significant screening ECG abnormality, or any other significant cardiovascular condition
* Presence of a gastrointestinal disease that could interfere with absorption of an orally administered drug
* Have epilepsy
* Positive urine drug test
* Prior adverse effects from psilocybin or other psychedelics that required hospitalization
* Currently taking on a regular basis (e.g., daily) any medications having a primary centrally acting serotonergic effect, including selective serotonin reuptake inhibitors (SSRIs), monoamine oxidase inhibitors (MAOIs), or serotonin-acting dietary supplements (such as 5-hydroxy-tryptophan or St. John's wort)
* Currently taking prohibited medications, including antihypertensive medications, UGT1A9 or 1A10 inhibitors (e.g., regorafenib, rifampicin, phenytoin, eltrombopag, mefenamic acid, diflunisal, niflumic acid, sorafenib, isavuconazole, deferasiroxor, ginseng), and aldehyde or alcohol dehydrogenase inhibitors (e.g,, disulfiram)
* Participation in another concurrent clinical study; or use of investigational drugs, biologics, or devices within 30 days prior to assignment of study drug administration order
* Anyone who is pregnant, lactating, or planning on becoming pregnant during the study
* Unwilling to withhold prohibited concomitant medications

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-06 (Estimated); Primary Completion 2024-03 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Determine the maximum concentration of psilocin following oral and IV administrations of psilocybin | Day 8, Day 22
  Determine the maximum plasma concentration of psilocin in plasma following a single IV dose as compared to that following a single oral dose.
Determine the concentration of psilocin following oral and IV administrations of psilocybin | Day 8, Day 22
  Determine the time to maximum plasma concentration of psilocin in plasma following a single IV dose as compared to that following a single oral dose.
Determine the concentration of psilocin following oral and IV administrations of psilocybin | Day 8, Day 22
  Determine the half-life of psilocin in plasma following a single IV dose as compared to that following a single oral dose.
Determine the concentration of psilocin following oral and IV administrations of psilocybin | Day 8, Day 22
  Determine the AUC of psilocin in plasma following a single IV dose as compared to that following a single oral dose.
Difference in the area under plasma concentration-time curve (AUC) between psilocybin administration methods. | Day 8, Day 22
  AUC will be determined after oral and IV psilocybin doses to assess for more consistent blood concentration.
Difference in the maximum concentration (Cmax) between psilocybin administration methods. | Day 8, Day 22
  Cmax will be determined after oral and IV psilocybin doses to assess for more consistent blood concentration.
Difference in the time to maximum plasma concentration (Tmax) between psilocybin administration methods. | Day 8, Day 22
  Tmax will be determined after oral and IV psilocybin doses to assess for more consistent blood concentration.

SECONDARY OUTCOMES:
Characterize the incidence and severity of adverse events associated with doses of psilocybin in healthy adults | 12 weeks
  The incidence and severity of expected and unexpected adverse events will be collected using the Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials
Suicidal ideation | 12 weeks
  Assessed using the Columbia - Suicide Severity Rating Scale (C-SSRS) at every in-person visit

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Nicholas, PhD, Principal Investigator — University of Wisconsin, Madison; Paul Hutson, PharmD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No